CLINICAL TRIAL: NCT05498376
Title: The Leadless AV Versus DDD Pacing Study: A Randomized Controlled Single-center Trial on Leadless Versus Conventional Cardiac Dual-chamber Pacing
Brief Title: The Leadless AV Versus DDD Pacing Study
Acronym: LEAVE DDD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-D0050
Record Dates: First submitted 2022-08-03; First posted 2022-08-12 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Pacemaker; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases
Keywords: Leadless pacemaker; Atrioventricular conduction block; Bradyarrhythmias; Micra
MeSH Terms: conditions — Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Atrioventricular Block; Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional pacemaker DDD (Active Comparator): Implantation of a conventional dual-chamber PM
  Interventions: Device: Conventional pacemaker DDD
- Leadless pacemaker Micra AV (Active Comparator): Implantation of a leadless pacemaker system (Micra AV™)
  Interventions: Device: Leadless pacemaker Micra AV

INTERVENTIONS:
Device: Conventional pacemaker DDD — Implantation of a conventional cardiac pacemaker
  Arms: Conventional pacemaker DDD
Device: Leadless pacemaker Micra AV — Implantation of a leadless cardiac pacemaker
  Arms: Leadless pacemaker Micra AV

SUMMARY:
Cardiac pacemaker (PM) implantation is the established treatment for relevant bradyarrhythmias. Conventional PMs require 1-3 pacing leads to register the heart's intrinsic activity ("sensing") and to deliver the electrical stimuli to the heart ("pacing"). These leads are responsible for the vast majority of morbidity after implantation and PM failures. Therefore, a leadless PM system (Micra TPS™, Medtronic, United States) has been introduced a few years ago. This system overcomes the limitations of leads, however, the first generation of the Micra TPS™ only allowed sensing and pacing in the right ventricle. More recently, an upgraded version has been introduced and gained market approval (Micra AV, Medtronic, United States). According to published results from several clinical trials, this device allows sensing the atrial activity and, thus, timing the delivery of the ventricular pacing impulse in a physiological manner similar to a conventional dual-chamber PM with two leads. Clinical feasibility and safety for this concept have been established already. However, it is unclear if this translates into a direct clinical benefit for patients in comparison to conventional PM systems.

The aim of this trial is to compare the therapeutic efficacy of the Micra AV™ PM and conventional dual-chamber PM systems in patients with intermittent or permanent atrioventricular conduction block and a PM indication according to the latest European guidelines. Thus, patients will be randomized to either a conventional dual-chamber PM implantation or the implantation of a leadless Micra AV™ system. Patients will be stratified for gender (female/male) and a priori estimated physical exercise capacity ("fit"/"unfit"). The primary outcome will be the physical exercise capacity of the patients.

The null hypothesis with regards to the primary endpoint is that the leadless pacemaker arm shows an inferior VO2 anaerobic threshold than the conventional pacemaker arm. Hence the alternative hypothesis postulates that the leadless pacemaker arm shows a non-inferior VO2 anaerobic threshold compared to the conventional pacemaker arm. Rejection of the null hypothesis is needed to conclude non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Patients (≥70y) undergoing a de-novo pacemaker implantation due to intermittent or permanent AV block, qualifying for a conventional or leadless pacemaker
* Written informed consent

Exclusion Criteria:

* Permanent atrial fibrillation or atrial standstill
* Evidence of sinus node disease and need for right atrial pacing (not possible with Micra AV)
* LVEF <50% and permanent high-degree or total AVB (requiring CRT/His-Bundle/CSP pacing)
* Preoperative E/A ratio >1.5 in the echocardiography
* Any co-existing ICD indications (no leadless ICD systems available)
* Hemodialysis
* Presence of a mechanical tricuspid valve prosthesis
* Unwilling or unable to comply fully with study procedures and follow-up

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity | Month 3 post implantation
  Exercise capacity (VO2 at anaerobic threshold) as assessed by spiroergometry

SECONDARY OUTCOMES:
Total implantation time | During implantation on day 0
  Total implantation time
Total fluoroscopy time | During implantation on day 0
  Total fluoroscopy time during implantation
Total fluoroscopy dosage | During implantation on day 0
  Total fluoroscopy dosage during implantation
Pacing thresholds | Days 0,1 and months 1,3,12 and 24 post implantation
  Pacing thresholds of the implanted pacemaker
Sensing values | Days 0,1 and months 1,3,12 and 24 post implantation
  Sensing values of the implanted pacemaker
Impedance values | Days 0,1 and months 1,3,12 and 24 post implantation
  Impedance values of the implanted pacemaker
Duration of exercise | Month 3 post implantation
  Duration of exercise until exhaustion assessed by spiroergometry
VO2max | Month 3 post implantation
  VO2max assessed by spiroergometry
VE/VCO2 | Month 3 post implantation
  VE/VCO2 assessed by spiroergometry
VE/VO2 | Month 3 post implantation
  VE/VO2 assessed by spiroergometry
Maximum atrial heart rate | Month 3 post implantation
  Maximum atrial heart rate as assessed by spiroergometry
Left ventricular ejection fraction (LVEF) | Day 0 and months 3, 12 and 24 post implantation
  LVEF as assessed by echocardiography
Degree of tricuspid valve regurgitation | Day 0 and months 3, 12 and 24 post implantation
  Degree of tricuspid valve regurgitation assessed by trans-thoracic echocardiogram. The degree of tricuspid valve regurgitation will be classified as "none", "mild", "moderate" or "severe"
Degree of mitral valve regurgitation | Day 0 and months 3, 12 and 24 post implantation
  Degree of mitral valve regurgitation assessed by trans-thoracic echocardiogram. The degree of mitral valve regurgitation will be classified as "none", "mild", "moderate" or "severe"
Quality of Life scores measured with the EQ-5D-5L Questionnaire | Days 0,1 and months 1,3,12 and 24 post implantation
  Quality of Life scores measured with the EQ-5D-5L Questionnaire Scores: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each with a 5-scale response option; current health state assessed with a number between 0 and 100
AV synchrony | Day 1 and months 1,3,12 and 24 post implantation
Laboratory | Day 0 and month 3 post implantation
  NT-proBNP
Safety outcomes | Days 0,1 and months 1,3,12 and 24 post implantation
  Major adverse events (death, cardiac tamponade, any surgical reintervention, pocket/groin problems, lead/device dislocations; electrode noise, pacing impedance out of range (<200 or >2000Ω), failure to capture at maximum output, infections and thrombosis/embolism); rate of pacemaker syndrome developed by patients; rate of device upgrades/revisions required

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Häberlin, MD, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Inselspital, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Brignole M, Auricchio A, Baron-Esquivias G, Bordachar P, Boriani G, Breithardt OA, Cleland J, Deharo JC, Delgado V, Elliott PM, Gorenek B, Israel CW, Leclercq C, Linde C, Mont L, Padeletti L, Sutton R, Vardas PE; ESC Committee for Practice Guidelines (CPG); Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Kirchhof P, Blomstrom-Lundqvist C, Badano LP, Aliyev F, Bansch D, Baumgartner H, Bsata W, Buser P, Charron P, Daubert JC, Dobreanu D, Faerestrand S, Hasdai D, Hoes AW, Le Heuzey JY, Mavrakis H, McDonagh T, Merino JL, Nawar MM, Nielsen JC, Pieske B, Poposka L, Ruschitzka F, Tendera M, Van Gelder IC, Wilson CM. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J. 2013 Aug;34(29):2281-329. doi: 10.1093/eurheartj/eht150. Epub 2013 Jun 24. No abstract available. PMID 23801822